CLINICAL TRIAL: NCT05373082
Title: Identification of Modifying Factors in Hereditary Spastic Paraplegia
Acronym: MODIFSPA2
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211621
Record Dates: First submitted 2022-03-04; First posted 2022-05-13 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hereditary spastic Paraplegia: Patients with hereditary spastic Paraplegia
  Interventions: Other: questionnaire completion

INTERVENTIONS:
Other: questionnaire completion — Questionnaire to be completed by patients

SUMMARY:
A first questionnaire - MODIFSPA conducted in 2014 - identified several environmental factors influencing spasticity in HSP: cold, fatigue, and especially physical activity. In order to improve the care of patients with HSP, The investigator team are looking to deepen the knowledge on physical exercises relieving spasticity as well as to better know the frequency of symptoms requiring additional medical care: fatigue and vesico-sphincter disorders. A new questionnaire was therefore created to collect additional information to optimize the care of patients with HSP.

DETAILED DESCRIPTION:
The only common symptom of hereditary spastic paraplegia (HSP) is the presence of spasticity in the lower limbs, associated with a great clinical and genetic heterogeneity.

A first MODIFSPA study carried out by the team identified environmental factors influencing spasticity: stress, fatigue, physical activity. In this first study, only spasticity was studied but several symptoms appeared to require medical management according to the patients: fatigue and vesico-sphincter disorders.

Following this first study, MODIFSPA2 aims to deepen our knowledge of HSP, via the expertise of patients, to propose a care in adequacy with their needs/demands.

Validated scales are included in the questionnaire to evaluate the frequency and intensity of the symptoms most reported by patients (fatigue, pain and mood disorders). Questions are asked to better know the frequency of symptoms requiring additional medical care: fatigue and vesico-sphincter disorders.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking adult patients aware of their PSH diagnosis coming to the genetic consultation at the Pitié-Salpêtrière Hospital or informed via an association / website of the BRAINTEAM study network
* Affiliated with social security

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Hereditary Spastic Paraplegia (HSP)
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
factors influencing spasticity | 1 day
  Temperature,stress, anxiety , intercurrent infection, physical activities and tiredness are the factors influencing spasticity (common symptom of all these patients): Only questions are asked with yes and no answers

SECONDARY OUTCOMES:
Physical activities | 1 day
  Does physical activity improve your health?
Symptoms | 1 day
  what symptoms do you have? fatigue, pain and vesico-sphincter disorders ( answers are yes or not)
Anxiety | 1 day
  Determine anxiety or depressive disorders (Hospital Anxiety and Depression scale; HAD) in this population anxiety max score>11 ( minimal anxiety score<7)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut du Cerveau, ICM, Paris, France